CLINICAL TRIAL: NCT03128710
Title: Identifying Patient-relevant Adverse Events Following Prostate Radiotherapy
Brief Title: Prostate Cancer Survey
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00073268
Record Dates: First submitted 2017-04-19; First posted 2017-04-25 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: Survey; Focus Group; Treatment Preferences
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survey Group: Approximately 300 patients with prostate cancer will be provided a survey investigating their treatment preferences and side effects faced during and after receiving radiation treatment.
- Focus Group: Approximately 75 participants will participate in a focus group. All participants will have completed radiation treatment and will discuss side effects after having received radiation, as well as their quality of life while receiving radiation.

SUMMARY:
There have been calls from patients, payers, healthcare providers, and policy makers for an evaluation of newer, high-cost radiation technologies compared to conventional forms of radiation therapy. National attention has focused on the use of intensity modulated radiation therapy (IMRT) into routine daily clinical practice for prostate cancer. The goal of the present study is to determine whether the type of radiation treatment received by the patients can result in a reduction in patient-relevant side effects following prostate irradiation. The analysis will be performed by obtaining patient answered surveys looking at side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years or older
* Has been diagnosed with prostate cancer
* Able to speak and read English

Exclusion Criteria:

* Participant is not being seen for prostate cancer
* Under the age of 18

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate malignancies who consent to receiving Radiation treatment at the University of Maryland, Baltimore, will be offered this survey.
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
To determine patient preference weights for side effect reduction in radiation treatment of prostate cancer | 3 years
  Investigators will use an anonymous survey and results from multiple focus groups to quantify the relative importance/significance of commonly encountered side effects experienced by patients following external beam radiation therapy. We will complete descriptive statistics as a means of understanding the data obtained by survey responses. Additionally, comparative analyses may be undertaken to evaluate differences between different side effects experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mishra, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- UMMC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No